CLINICAL TRIAL: NCT06040203
Title: Leukocyte-rich PRP or Leukocyte-free PRP vs Placebo in the Treatment of Epicondylitis: a Randomized Controlled Clinical Trial
Brief Title: Leukocyte-rich PRP or Leukocyte-free PRP vs Placebo in the Treatment of Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Epic-PRP
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Tennis Elbow
Keywords: Platelet rich plasma; Leukocyte-rich PRP; Leukocyte-poor PRP; PRP; PRP injection; Double-blind randomized controlled clinical trial
MeSH Terms: conditions — Tennis Elbow | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomized controlled clinical trial with 1:1:1 allocation
Who Masked: Participant, Outcomes Assessor
Masking Description: They will be "blinded" patients, health professionals who will assess clinical and functional outcomes (outcome assessors), and professionals who will analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leukocyte-rich Platelet rich plasma (LR-PRP) (Experimental): This group of patients will be treated with single injection of autologous leukocyte rich platelet rich plasma.At the 6-month follow-up visit, the patient will be informed about the treatment received.
  Interventions: Biological: Injection of autologous leukocyte rich platelet rich plasma (LR-PRP)
- Leukocyte-poor Platelet rich plasma (LP-PRP) (Experimental): This group of patients will be treated withsSingle injection of autologous leukocyte poor platelet rich plasma.At the 6-month follow-up visit, the patient will be informed about the treatment received.
  Interventions: Biological: Injection of autologous leukocyte poor platelet rich plasma (LP-PRP)
- Saline solution (Placebo Comparator): This group of patients will be treated with single intra-articular injection of saline solution (placebo). At the 6-month follow-up visit, patients will be informed about the treatment received. Patients of this group can cross-over to the treatment arm after 6 months following a dedicated randomization list.
  Interventions: Drug: Placebo (saline solution)

INTERVENTIONS:
Biological: Injection of autologous leukocyte rich platelet rich plasma (LR-PRP) — Patients will be treated with a single eco-guided injection of Autologous LR-PRP in the elbow affected by epicondylitis.
  Arms: Leukocyte-rich Platelet rich plasma (LR-PRP)
Biological: Injection of autologous leukocyte poor platelet rich plasma (LP-PRP) — Patients will be treated with a single eco-guided injection of Autologous LP-PRP in the elbow affected by epicondylitis.
  Arms: Leukocyte-poor Platelet rich plasma (LP-PRP)
Drug: Placebo (saline solution) — Patients will be treated with a single injections of saline solution in the elbow affected by epicondylitis.
  Arms: Saline solution

SUMMARY:
The EPIC-PRP study is a double-blind randomized controlled clinical trial with 1:1:1 allocation.The objective of the study is to evaluate by means of a randomized controlled, double-blind clinical trial the clinical outcomes of echo-guided injection of PRP with or without leukocytes compared with echo-guided injection of saline for minimally invasive treatment of patients with epicondylitis resistant to conservative therapy. It will be the aim of the study to evaluate the efficacy and safety of the injection procedures by revealing the improvement and incidence of adverse events following treatment

DETAILED DESCRIPTION:
Patients with elbow epicondylitis will be included in a double-blind, randomized controlled trial, in which one group of patients will be treated with an echo-guided injection of LP-PRP (low leukocyte PRP), one group of patients will be treated with an echo-guided injection of LR-PRP (high leukocyte PRP), and another group of patients will be treated with an echo-guided injection of saline.All enrolled patients undergo sampling of a venous whole blood bag of approximately 300 cc from which Fresh Autologous PRP (PRP-A) will subsequently be obtained. According to randomization, a "leukodepletion" filter will be used to remove leukocytes in order to obtain LP-PRP. Instead, an aliquot of PRP will be cryopreserved and made available for the patient for a possible second PRP infiltration if there is no benefit after 6 months after the first infiltration.The patient will then be placed on the randomization list and will, therefore, be assigned to one of the three treatment groups (leukocyte-rich PRP, leukocyte-poor PRP, or saline solution). In the case of patients in the saline injection group, PRP will be prepared with or without leukocytes according to a dedicated randomization list, for possible treatment after 6 months if necessary.The patient will subsequently undergo 1 echo-guided infiltration, according to randomization.Patients will be clinically evaluated before the infiltration procedure and at 1-3-6-12 months after treatment by medical personnel. Questionnaires will be administered for clinical evaluations before treatment and at the above-mentioned clinical checkups during follow-up. Any adverse events to treatment will also be evaluated during follow-up visits. The duration and extent of swelling and pain following infiltration will be reported, and any drug therapies given by the patient will be recorded

ELIGIBILITY:
Inclusion Criteria:

Patients with epicondylitis of the elbow:

1. Patients with clinical picture of epicondylitis;
2. Duration of symptoms > 3 months
3. Ultrasound picture of short or long radial extensor carpal tendinopathy;
4. Age > 18 and < 65
5. Both sexes;
6. Failure, defined as persistence of symptoms, of other conservative treatments for at least 3 months;
7. Hemoglobin > 11 g/dl;
8. Platelet count > 150,000 plt/mm3 (Recently performed CBC examination);
9. Negative serological tests for HBsAg, HCV Ab, HIV-1-2 Ab
10. No clinically significant electrocardiographic changes (Recently performed ECG);
11. Ability and consent of the patient to actively participate in clinical follow-up;
12. Signature of informed consent.

Exclusion Criteria:

1. Patients undergoing previous surgical treatment on the epicondylar tendons;
2. Patients undergoing epicondylar infiltration in the previous 6 months;
3. Inability of patients to actively participate in clinical follow-up;
4. Incapacitated patients;
5. Patients with states of immunodepression;
6. Patients with fibromyalgia;
7. Ongoing systemic inflammatory diseases (stabilized outcomes of such diseases are not considered absolute contraindications);
8. Patients with uncontrolled thyroid metabolic disorders;
9. Patients abusing alcoholic beverages, drugs or medications;
10. Patients who have taken NSAIDs in the 3 days prior to blood collection;
11. Patients with coagulation problems or with ongoing antiplatelet therapy that cannot be suspended for at least 3 days prior to blood draw;
12. Patients with cardiovascular disease for whom a 300-mL blood draw would be contraindicated;
13. Positive serological tests for HBsAg, HCV Ab, HIV-1-2 Ab
14. Other current elbow diseases (osteoarthritis, prevalence of symptomatology due to epitrochleitis, stiff elbow, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Patient-rated Tennis Elbow Evaluation (PRTEE) | 6 months follow-up
  PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis (also known as "tennis elbow"). The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales: 1) Pain subscale (0 = no pain, 10 = worst imaginable) item 2) Function subscale (0 = no difficulty, 10 = unable to do).
  The total score is the sum of the two subscales and has a range from 0 to 100.

SECONDARY OUTCOMES:
Patient-rated Tennis Elbow Evaluation (PRTEE) | baseline, 1 month, 3 months and 12 months follow-up
  PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis (also known as "tennis elbow"). The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales: 1) Pain subscale (0 = no pain, 10 = worst imaginable) item 2) Function subscale (0 = no difficulty, 10 = unable to do).
  The total score is the sum of the two subscales and has a range from 0 to 100.
Disability of the arm, shoulder and hand score (DASH) | baseline, 1 month, 3 months, 6 months and 12 months follow-up
  The Disabilities of the Arm, Shoulder and Hand (DASH) Score is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Tegner Activity Level Scale | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Tegner Activity Level Scale is a questionnaire to find out the patient's level of physical activity.All patients will indicate the type of sporting activity performed and its frequency.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability and 10 represents a competitive level of sport.
Oxford Elbow Score (OES) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Oxford Elbow score is a questionnaire consisting of 12 questions (related to pain, function, and socio-psychological aspects) specifically designed and developed to evaluate the outcomes of elbow surgery.
  The Oxford Elbow score has 12 items (questions) with 5 response options each. Each item response is scored as 0 to 4, with 0 representing greater severity. Underlying the 12 items are 3 domains (subscales): elbow pain, elbow function and social-psychological effects. Scores for each domain are calculated as the sum of each individual item score within that domain. This gives a score range of 0-16 for each domain and 0-48 overall, with 0 indicating the worst elbow score and 48 as a 'normal' elbow score
Visual Analogue Scale (VAS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" (0) and "the strongest pain imaginable" (10).
EuroQol Visual Analogue Scale (EQ-VAS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  EQ-VAS is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
EQ-5D (EuroQoL) Current Health Assessment | baseline, 1 month, 3 months, 6 and 12 months follow-up
  The generic health-related quality of life instrument-EQ-5D-allows both a description of health status along 5 dimensions and the evaluation of health or the estimation of a health summary score: the EQ-5D score on a scale where 0 is death and 1 is full health. EQ-5D is useful to evaluate the quality life of the patients. The EQ-5D respondents classify their own health status into 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with 3 levels of severity (no problems, moderate problems, or severe problems).
Pain detect | baseline
  The Pain Detect-Questionnaire is a reliable screening tool for neuropathic pain with high sensitivity, specificity, and positive predictive accuracy. In this scale, the score ranges from 0 to 38 (range 0-12 neuropathic component of pain unlikely, range 13-18 neuropathic component of pain probably present, range 19-38 neuropathic component of pain present).
Patient Acceptable Symptom State (PASS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Final treatment opinion | 1 month, 3 months, 6 and 12 months follow-up
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
Effectiveness of the blinding procedure | baseline
  The patient should indicate, after the infiltrative procedure, the type of treatment they think they received.
Expectations of treatment efficacy | baseline
  The patient should indicate at baseline what benefits they expect from the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Guerra, MD, Principal Investigator — Istituto Ortopedico Rizzoli - SC Chirurgia della spalla e del gomito
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Kim GM, Yoo SJ, Choi S, Park YG. Current Trends for Treating Lateral Epicondylitis. Clin Shoulder Elb. 2019 Dec 1;22(4):227-234. doi: 10.5397/cise.2019.22.4.227. eCollection 2019 Dec. PMID 33330224
- [Background] Chen J, Wang A, Xu J, Zheng M. In chronic lateral epicondylitis, apoptosis and autophagic cell death occur in the extensor carpi radialis brevis tendon. J Shoulder Elbow Surg. 2010 Apr;19(3):355-62. doi: 10.1016/j.jse.2009.07.064. PMID 19836974
- [Background] Hsu WK, Mishra A, Rodeo SR, Fu F, Terry MA, Randelli P, Canale ST, Kelly FB. Platelet-rich plasma in orthopaedic applications: evidence-based recommendations for treatment. J Am Acad Orthop Surg. 2013 Dec;21(12):739-48. doi: 10.5435/JAAOS-21-12-739. PMID 24292930
- [Background] Chen X, Jones IA, Park C, Vangsness CT Jr. The Efficacy of Platelet-Rich Plasma on Tendon and Ligament Healing: A Systematic Review and Meta-analysis With Bias Assessment. Am J Sports Med. 2018 Jul;46(8):2020-2032. doi: 10.1177/0363546517743746. Epub 2017 Dec 21. PMID 29268037
- [Background] Karaduman M, Okkaoglu MC, Sesen H, Taskesen A, Ozdemir M, Altay M. Platelet-rich plasma versus open surgical release in chronic tennis elbow: A retrospective comparative study. J Orthop. 2016 Jan 22;13(1):10-4. doi: 10.1016/j.jor.2015.12.005. eCollection 2016 Mar. PMID 26955228